CLINICAL TRIAL: NCT06584266
Title: Multimodal, Multicentre Registry of Clinical and Imaging Data to Develop Predictive Models Based on Artificial Intelligence to Support the Diagnostic and Therapeutic Process for Patients with Atrial Fibrillation Undergoing Catheter Ablation and Cardioversion.
Brief Title: Multimodal Cardiac Imaging Registry in Patients with Atrial Fibrillation
Acronym: IMAGE-AF
Status: Recruiting | Type: Observational
Sponsor: University in Zielona Góra (Other)
Collaborators: Military Institute od Medicine National Research Institute (Other); National Institute of Cardiology, Warsaw, Poland (Other); Medical University of Silesia, Katowice, Poland (Unknown); St. Anne's University Hospital Brno, Czech Republic (Other); John Paul II Hospital, Krakow (Other); Nowa Sol Multidyscyplinary Hospital, Poland (Unknown)
Responsible Party: Principal Investigator, Konrad Pieszko, MD, PhD, University in Zielona Góra
Other Study IDs: 1/KARD/UZ/2023
Record Dates: First submitted 2024-08-31; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation and Flutter; Heart Failure; Artificial Intelligence (AI); Echocardiography
Keywords: artificial intelligence; left atrial thrombus; transesophageal echocardiography; left atrial appendage thrombus; ablation; left atrial function
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Echocardiography, Transesophageal; Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AF or AFl patients: Patients with AF or AFl in whom TEE will be performed (to assess their eligibility for cardioversion or ablation), hospitalized in a participating center during study period.
  Interventions: Diagnostic Test: Transoesophageal echocardiography; Procedure: Catheter ablation

INTERVENTIONS:
Diagnostic Test: Transoesophageal echocardiography — Imaging data obtained with transoesophageals echocardiography will be retained as well as data from transthoracic echocardiography and from other imaging modalities, if available
Procedure: Catheter ablation — Cathether ablation of atrial fibrillation substrate using one of available methods.

SUMMARY:
The goal of this observational registry is to collect a curated dataset of multimodal imaging data that will serve for development of artificial-intelligence based solutions for prediction of risk and outcomes in patients with atrial fribrillation.

Type of study: observational study

Study Participants: Patients with atrial fibrillation or atrial flutter who undergo clinically indicated transesophageal echocardiography before catheter ablation or cardioversion.

We hypothesize, that automatic analysis of video images of transthoracic echocardiography with deep learning combined with clinical data can predict the presence of left atrial appendage thrombus (LAT). Therefore, our main aim is to create and validate an artificial intelligence model to predict the presence of LAT based on automatic analysis of transthoracic echocardiography with artificial intelligence.

DETAILED DESCRIPTION:
1. Introduction

   Atrial fibrillation (AF) is the most common cardiac arrythmia, that affects 37% Europeans over 55 years old, representing a major burden for the society and health systems. One of the most devastating consequences of AF is ischemic stroke, often caused by embolization of cerebral arteries with a left atrial appendage thrombus (LAT), which can form in left atrial appendage in the presence of AF. As it has little contractility on its own, emptying and filling of left atrial appendage relies on the function of the left ventricle and the left atrium.

   AF as well as atrial flutter promote the formation of LAT and are therefore associated with an increased risk of thromboembolic events. The mechanism of stroke is complex, but embolization with LAT accounts for the majority of events and it can be triggered by sinus rhythm restoration through procedures commonly performed in patients with AF - cardioversion or catheter ablation. Therefore, cardioversion and catheter ablation in the presence of LAT are contraindicated.

   Transoesophageal echocardiography (TEE) is considered the modality of choice to detect LAT with high sensitivity and specificity and is currently recommended before cardioversion or catheter ablation as an alternative to a 3-week course of oral anticoagulation. Current guidelines, however, leave room for an individual decision to either perform or not perform TEE before catheter ablation or cardioversion in a chronically anticoagulated patient but suggest no tools to assess the risk of LAT. To address this unmet clinical need, we have previously shown that by combining clinical data and measurements from transthoracic echocardiography in a machine-learning model it is possible to predict the risk of LAT formation. Importantly, our results indicated, that TTE-derived measurements played the greatest role in predicting LAT.

   Despite significant advancements in interventional technologies, the selection of appropriate therapeutic methods and perioperative procedures remains a significant challenge. Patients eligible for interventional procedures related to AF often undergo numerous diagnostic tests, including computed tomography of the heart, transoesophageal and transthoracic echocardiography, electrocardiography (EKG), and electroanatomic mapping during the ablation procedure. Non-invasive multimodal imaging plays central role in the peri-ablation period, informing important therapeutic decisions and facilitating the procedure. The essence of this project is the prospective collection of high-quality imaging data from these multiple modalities and clinical data, which will allow for a better understanding of the relationships between anatomy, hemodynamic function, and clinical observation in patients with AF in the future. Ultimately the data might serve for the development of tools which could efficiently predict the risk of LAT by means of less invasive and cheaper approaches than the ones which are currently used. The resulting multimodal database will also form a foundation for future studies targeted at informing therapeutic decisions in patients undergoing catheter ablation of AF.
2. Study Objectives

   2.1. Main objective: To create a multimodal, multicentre registry of clinical and imaging data to develop predictive models based on state-of the art artificial intelligence to support the diagnostic and therapeutic process for patients undergoing AF catheter ablation and cardioversion.

   2.2. Specific objectives:

   2.2.1. Specific Aim 1 Creation of artificial intelligence-based models to predict the risk of formation of left atrial appendage thrombus and estimate the left atrial appendage emptying velocity obtained from transoesophageal echocardiography based on the analysis of transthoracic echocardiographic images and clinical data.

   2.2.2. Specific Aim 2 Assessment of inter-reader and intra-reader agreement in the clinical interpretation of left atrial appendage images and left atrial appendage thrombus diagnosis in transoesophageal echocardiography.

   2.2.3. Specific Aim 3 Development of models that fuse information from multiple modalities (for instance from transthoracic echocardiography and cardiac CT) to provide better prognosis and guide therapeutic decisions in patients with atrial fibrillation.

   2.2.4. Specific Aim 4 Comparison of the effectiveness of different methods of imaging the left atrium in predicting thromboembolic events.

   2.2.5. Specific Aim 5 Creation of a high-quality multicentre imaging database for additional future auxillary nalyses and studies.
3. Study Methodology

   To maximize the amount of collected data the study allows both retrospective and prospective data collection. The scope of collected data is the same in retrospective and prospective collection with certain data types being optional and subject to availability.

   3.1. Inclusion criteria

   Patients with:
   * history of atrial fibrillation,
   * who are undergoing medically justified transoesophageal echocardiography to assess the presence of left atrial appendage thrombus before catheter ablation of atrial fibrillation (including patients who had transoesophageal echocardiography during the ablation procedure). OR
   * who undergo catheter ablation without prior transoesophageal echocardiography (if the center also collects additional imaging data listed in point 2.5 below) 3.2. Exclusion criteria
   * Age < 18 years old.

   3.3 3.3. Types of collected data

   Data type: Clinical data Compulsory or optional: Includes compulsory and optional fields Format: Tabular, collected using a dedicated eCRF Additional remarks: The detailed list of fields with possible values is shown in Appendix 1

   Data type: TTE Compulsory or optional: Compulsory Format: DICOM Additional remarks: Recorded before TEE preferably on the same day. In case of retrospective data TTE and TEE acquired within 72h

   Data type: TEE Compulsory or optional: Compulsory if the patient had TEE Format: DICOM

   Additional remarks:

   Data type: Cardiac CT Compulsory or optional: Optional Format: DICOM Additional remarks: Contrast enhanced cardiac CT before ablation procedure. Can be a study performed for EP planning or for CAD diagnostics. Any study performed before the ablation regardless of timing can be used

   Data type: Non-contrast Cardiac CT Compulsory or optional: Optional Format: DICOM Additional remarks: Non-contrast chest CT. Preferred is ECG-gated calcium scoring CT reconstructed with thin slices (preferably 0.5mm).

   Data type: Cardiac Magnetic Resonance (CMR) Compulsory or optional: Optional Format: DICOM

   Additional remarks:

   Data type: Digitalised Electrocardiogram Compulsory or optional: Optional Format: DICOM (or pdf) Additional remarks: Performed on the day of the catheter ablation or cardioversion or day before.

   Data type: Electroanatomical map Compulsory or optional: Optional Format: Proprietary Additional remarks: Not to be transferred but only stored locally in the participating center for possible ancillary studies

   Data type: Follow-up for MACE Compulsory or optional: Optional Format: Event date Additional remarks: Depending on the local regulations and possibility, the follow-up data for all-cause mortality, stroke, myocardial infarction, onset or worsening of heart failure will be obtained based on ICD-9 and ICD 10 codes from the national health insurance databases. Alternatively, data can be obtained by telephone interview

   Data type: Follow-up for AF Compulsory or optional: Optional Format: Event date Additional remarks: Depending on the local availability of follow-up data for AF recurrence

   3.4. Guidelines for data acquisition

   3.4.1. Guidelines for Acquisition of Transthoracic and Transesophageal Echocardiography
   * For prospective collection the TEE and TEE should be performed ideally in the same day, TTE directly before TEE. For the retrospective cohort TTE can be acquired up to 3 days before TEE, as long as there were no important changes in patients' condition during this period (i.e. clinical worsening, change of rhythm, heart rate etc).
   * ECG electrodes should be connected for both TTE and TEE (not compulsory for retrospective data)
   * The acquisition length should be set to 5 seconds (set the start acquisition at the moment when acquire button is pressed to minimise unwanted movement). For retrospective data shorter clips are acceptable.

   3.4.1.1. Acquisition of TTE [filenames are given in brackets]:
   1. Four-chamber apical projection [4ch.dcm]
   2. Two-chamber apical projection [2ch.dcm]
   3. Three-chamber apical projection [3ch.dcm]
   4. Four-chamber apical projection - optimized for LA [4chLA.dcm]
   5. Two-chamber apical projection - optimized for LA [2chLA.dcm]
   6. 3D full volume (preferably acquired from 4 or more heart cycles) [3d_tte.dcm] The projections must encompass the entire heart, including the atria. Measurements to be performed at site (if impossible, some of these measurements can also be performed by the coordinating site).

   <!-- -->

   1. Cardiac chamber dimensions (PLAX) [plax.dcm]
   2. Velocities E, A, med. E', lat. E' (still images) [mitral_flow.dcm, medial_tdi.dcm, lateral_tdi.dcm]
   3. Tricupid regurgitation spectral image (still images) [tr.dcm]

   3.4.1.2. Acquisition of TEE:
   1. Projection on LAA (Left Atrial Appendage): 0, 45, 90, 135 degrees, and other projections that are necessary to correctly image the entire LAA according to the investigator/ echocardiographer [laa_0.dcm, laa_45.dcm, laa_135.dcm etc.]
   2. 3D acquisition of the volume that contains LAA (multi-beat-optimized) [3d_LAA.dcm]
   3. Measurement of maximum emptying velocity of LAA 1cm from the LAA ostium - at least three measurements in two different scanning angles, averaged.
   4. Acquisition of spectral Doppler image of LAA emptying (three images from two or more scanning angles) (still images) [laav_60.dcm, laav135.dcm, laav_45.dcm]

      3.4.1.3. Other modalities: There are no specific acquisition requirements for cardiac CT, CMR or ECG - these studies should be performed according to local standard protocols.

      Appendix 1 - Dictionary of tabular data

      Variable: CaseID Display name: Case ID Type: ID Compulsory: Yes Categories and Units details: Consecutive IDs unique for each entry

      Variable: PatientID Display name: Patient ID Type: ID Compulsory: Yes Categories and Units details: Consecutive ID for patients; if the patient is entered to the registry more than once, he/she should have the same PatientID

      Variable: procedure_type Display name: Type of planned intervention Type: Clinical Compulsory: Yes Categories and Units details: ablation = 1, cardioversion = 2, NA = 3, laa_closure = 4, valvular disease = 5, infective endocarditis = 6

      Variable: AF Display name: Atrial fibrillation Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: AFL Display name: Atrial flutter Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: arrythmia_duration Display name: Paroxysmal, persistent, or long-standing Type: Clinical Compulsory: Yes Categories and Units details: persistent = 1, paroxysmal = 2, long-standing persistent = 3, NA = 4

      Variable: Persistent_arrythmia_time Display name: Time since the onset of persistent arrythmia Type: Clinical Compulsory: Yes Categories and Units details: Time in months or days. Enter 0 for paroxysmal arrythmia

      Variable: Persistent_arrythmia_time_unit Display name: Months or days Type: Clinical Compulsory: Yes Categories and Units details: Months = 0, Days = 1

      Variable: Disease_duration Display name: Duration of AF Disease Type: Clinical Compulsory: Yes Categories and Units details: Time (approximate) since the first diagnosis of atrial fibrillation

      Variable: Disease_duration_unit Display name: Months or Years Type: Clinical Compulsory: Yes Categories and Units details: Months = 0, Years = 1

      Variable: EHRA Display name: EHRA scale Type: Clinical Compulsory: Yes Categories and Units details: I = 1, IIa = 2, IIb = 3, III = 4, IV = 5, NA = 6

      Variable: Age Display name: Age Type: Clinical Compulsory: Yes Categories and Units details: Age in years

      Variable: Sex Display name: Sex Type: Clinical Compulsory: Yes Categories and Units details: Male = 1, Female = 2

      Variable: Height Display name: Height Type: Clinical Compulsory: Yes Categories and Units details: Height in cm

      Variable: Weight Display name: Weight Type: Clinical Compulsory: Yes Categories and Units details: Weight in kg

      Variable: HF_status Display name: Heart failure Type: Clinical Compulsory: Yes Categories and Units details: HFmrEF= 1, HFpEF = 2, HFrEF = 3, No HF = 4

      Variable: NYHA Display name: NYHA scale Type: Clinical Compulsory: Yes Categories and Units details: I = 0, II = 1, III = 2, IV = 3, No HF = 4

      Variable: MS Display name: Mitral stenosis Type: Clinical Compulsory: Yes Categories and Units details: mild = 1, moderate = 2, severe = 3, no MS = 4

      Variable: MR Display name: Mitral regurgitation Type: Clinical Compulsory: Yes Categories and Units details: mild = 1, moderate = 2, severe = 3, no MR = 4

      Variable: AS Display name: Aortic stenosis Type: Clinical Compulsory: Yes Categories and Units details: mild = 1, moderate = 2, severe = 3, no AS = 4

      Variable: AR Display name: Aortic regurgitation Type: Clinical Compulsory: Yes Categories and Units details: mild = 1, moderate = 2, severe = 3, no AR = 4

      Variable: mitral_valve_replacement Display name: Mitral valve replacement Type: Clinical Compulsory: Yes Categories and Units details: biological = 1, mechanical = 2, No MVR = 3

      Variable: aortic_valve_replacement Display name: Aortic valve replacement Type: Clinical Compulsory: Yes Categories and Units details: biological = 1, mechanical = 2, No AVR = 3

      Variable: Implanatable_device Display name: Presence of implantable electronic device Type: Clinical Compulsory: Yes Categories and Units details: None = 0, pacemaker = 1, ICD = 2, CRT-D = 3, CRT-P = 4, Implantable Recorder = 5, S-ICD = 6, Leadless pacemaker = 7

      Variable: stroke_type Display name: History of stroke Type: Clinical Compulsory: Yes Categories and Units details: haemorrhagic stroke = 1, ischaemic stroke = 2, both = 3, no history of stroke = 4

      Variable: peripheral_embolus Display name: History of peripheral embolism Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: revasc Display name: Prior revascularisation Type: Clinical Compulsory: Yes Categories and Units details: CABG = 1, No history of revasc = 2, PCI = 3, PCI+CABG = 4

      Variable: cad Display name: Coronary Artery Disease Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: vascular_disease Display name: Vascular disease Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: past_bleeding Display name: History of bleeding Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: CKD Display name: Chronic kidney disease Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: HT Display name: Hypertension Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: DM Display name: Diabetes Mellitus Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: liver_disease Display name: Liver disease Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: labile_INR Display name: Labile INR Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: alcohol Display name: Alcohol abuse Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: smoking Display name: Smoking Type: Clinical Compulsory: Yes Categories and Units details: currently = 1, in the past = 2, non-smoker = 3

      Variable: malignant_tumor Display name: Malignant tumor or cancer Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0, Malignant tumor or cancer or hematologic malignant disease

      Variable: COPD Display name: Chronic obstructive pulmonary disease Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: asthma Display name: Asthma Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: hyperthyroidism Display name: Hyperthyroidism Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: hypothyroidism Display name: Hypothyroidism Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: LA_dimension Display name: Left atrial AP dimension Type: TTE Compulsory: Yes Categories and Units details: Value in mm

      Variable: LVDd Display name: Left ventricular internal diameter end diastole Type: TTE Compulsory: Yes Categories and Units details: Value in mm

      Variable: RVDd Display name: Right ventricular internal diameter end diastole Type: TTE Compulsory: Yes Categories and Units details: Value in mm

      Variable: EF_TTE Display name: Left Ventricular Ejection Fraction Type: TTE Compulsory: Yes Categories and Units details: Value in %

      Variable: LA_area_4ch Display name: Left atrial area in four-chamber view Type: TTE Compulsory: Yes Categories and Units details: Value in cm2

      Variable: LA_length_4ch Display name: Left atrial length in four-chamber view Type: TTE Compulsory: No Categories and Units details: Value in cm

      Variable: LA_area_2ch Display name: Left atrial area in two-chamber view Type: TTE Compulsory: No Categories and Units details: Value in cm2

      Variable: LA_length_2ch Display name: Left atrial length in two-chamber view Type: TTE Compulsory: No Categories and Units details: Value in cm

      Variable: LA_volume_sp Display name: Left atrial single-plane volume Type: TTE Compulsory: No Categories and Units details: Value in cm3

      Variable: LA_volume Display name: Left atrial biplane volume Type: TTE Compulsory: No Categories and Units details: Value in cm3

      Variable: LAVI Display name: Left atrial volume index Type: TTE Compulsory: No Categories and Units details: Value in cm3/m2

      Variable: E Display name: Peak E-wave velocity Type: TTE Compulsory: Yes Categories and Units details: Value in cm/s

      Variable: A Display name: Peak A-wave velocity Type: TTE Compulsory: Yes Categories and Units details: Value in cm/s

      Variable: Med_Eprim Display name: Med E' - Early diastolic medial mitral annulus velocity Type: TTE Compulsory: Yes Categories and Units details: Value in cm/s

      Variable: Lat_Eprim Display name: Lat E' - Early diastolic lateral mitral annulus velocity Type: TTE Compulsory: Yes Categories and Units details: Value in cm/s

      Variable: RA area Display name: Right atrial area Type: TTE Compulsory: No Categories and Units details: Value in cm2

      Variable: Act Display name: Pulmonary acceleration time Type: TTE Compulsory: Yes Categories and Units details: Value in ms

      Variable: lab_date Display name: Lab Test Date Type: Lab Tests Compulsory: No Categories and Units details: If blood sample was drawn during hospitalization and lab test results are entered, please provide the date of lab tests

      Variable: BNP Display name: NT-proBNP Type: Lab Tests Compulsory: No

      Categories and Units details:

      Variable: Fib Display name: Fibrynogen Type: Lab Tests Compulsory: No

      Categories and Units details:

      Variable: CRP Display name: C-reactive Protein Type: Lab Tests Compulsory: No

      Categories and Units details:

      Variable: APTT Display name: Activated partial Thromboplastin Time Type: Lab Tests Compulsory: No

      Categories and Units details:

      Variable: INR Display name: International Normalized Ratio Type: Lab Tests Compulsory: No

      Categories and Units details:

      Variable: Hb Display name: Hemoglobin Type: Lab Tests Compulsory: No

      Categories and Units details:

      Variable: RDW Display name: Red Cell Distribution Width Type: Lab Tests Compulsory: No

      Categories and Units details:

      Variable: Crea Display name: Creatinine Type: Lab Tests Compulsory: No Categories and Units details: mg/dl

      Variable: months_anticoagulation Display name: Months since initiation of anticoagulation Type: Medication Compulsory: Yes Categories and Units details: Time in months; if more than one year, enter 12

      Variable: days_anticoagulation Display name: Days since initiation of anticoagulation Type: Medication Compulsory: Yes Categories and Units details: (if <1 month, otherwise leave blank)

      Variable: anticoagulant Display name: Type of anticoagulant medication Type: Medication Compulsory: Yes Categories and Units details: apixaban_2x5 = 1, rivaroxaban_20 = 2, dabigatran_2x150 = 3, acenocumarol = 4, warfarin = 5, apixaban_2x2.5 = 6, rivaroxaban_15 = 7, dabigatran_2x110 = 8, LVH = 9, HNF = 10, no anticoagulation = 11

      Variable: days_dabigatran_temp_use Display name: Temporary use of dabigatran (days) Type: Medication Compulsory: Yes Categories and Units details: Explanation: This is perhaps site-specific. In our center, we change medication to dabigatran in the periprocedural period because of access to praxbind.

      Variable: ASA Display name: intake of acetylsalicylic acid Type: Medication Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: clopidogrel Display name: intake of clopidogrel Type: Medication Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: tikagrelor Display name: intake of tikagrelor Type: Medication Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: prasugrel Display name: intake of prasugrel Type: Medication Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: base_rythm Display name: Rhythm at the time of study Type: Clinical Compulsory: Yes Categories and Units details: SR = 1, AF = 1, Afl = 2

      Variable: TEE_in_cath_lab Display name: TEE performed in cath lab Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0; indicates if TEE was performed during the ablation procedure

      Variable: TEE_historyof_LAT Display name: History of LAT in TEE Type: Clinical Compulsory: Yes Categories and Units details: Yes = 1, No = 0; indicates that the patient had TEE in the past where LAT was present

      Variable: TEE_historyof_LAT_date Display name: Date of TEE where LAT was diagnosed in the past Type: Clinical Compulsory: No Categories and Units details: If above is true, provide date of previous TEE

      Variable: TEE_SEC Display name: transesophageal echocardiography spontaneous echo contrast Type: TEE Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: TEE_DSEC Display name: transesophageal echocardiography dense spontaneous echo contrast Type: TEE Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: TEE_LAAV Display name: transesophageal echocardiography left atrial appendage flow velocity Type: TEE Compulsory: Yes Categories and Units details: value in cm/s

      Variable: TEE_LAT Display name: Presence of left atrial appendage thrombus Type: TEE Compulsory: Yes

      Categories and Units details:

      Variable: CT_date Display name: Date of computed tomography Type: Other modalities Compulsory: No Categories and Units details: If CT was performed, date of scan

      Variable: CT_DICOM_available Display name: Availability of CT DICOM data Type: Other modalities Compulsory: Yes Categories and Units details: Yes = 1, No = 0

      Variable: CT_CAC_score Display name: Coronary Artery Calcium Score Type: Other modalities Compulsory: No Categories and Units details: If CAC scan was performed, CAC score in Agatston Units

      Variable: CT_LA_Volume Display name: LA Volume in CT Type: Other modalities Compulsory: No Categories and Units details: ml; only if LA volume was assessed in CT

      Variable: ECG_date Display name: Date of ECG Type: Other modalities Compulsory: No

      Categories and Units details:

      Variable: ECG_dicom_available Display name: Availability of ECG DICOM data Type: Other modalities Compulsory: No

      Categories and Units details:

      Variable: CMR_date Display name: Date of Cardiac Magnetic Resonance Type: Other modalities Compulsory: No

      Categories and Units details:

      Variable: CMR_dicom_available Display name: Availability of CMR DICOM data Type: Other modalities Compulsory: No

      Categories and Units details:

      Variable: ablation_type Display name: Type of catheter ablation Type: Ablation Compulsory: No Categories and Units details: Cryobaloon ablation = 1, Pulsed field ablation = 2, RF ablation = 3, Other = 4

      Variable: first_ablation Display name: First ablation or re-do Type: Ablation Compulsory: No Categories and Units details: Yes = 1, No = 0 (0 indicates re-do)

      Variable: electroanatomical_mapping Display name: Type of catheter ablation Type: Ablation Compulsory: No Categories and Units details: Yes = 1, No = 0; indicates if the procedure was electroanatomical map was created

      Variable: LVZ Display name: Presence of low-voltage zones (LVZ) Type: Ablation Compulsory: No Categories and Units details: Yes = 1, No = 0; LVZ should be measured in sinus rhythm excluding pulmonary veins, preferably with multipolar catheter. Threshold: <0.5mV on sinus rhythm, <0.3mV on AF

      Variable: LVZ_locations Display name: Locations of LVZ Type: Ablation Compulsory: No Categories and Units details: Multiple choice: anterior wall, posterior wall, superior wall (Huo T., Gaspar M., Pohl et al. Europace 20 (2018) 956-962)

      Variable: ablation targets Display name: Regions of ablation energy Type: Ablation Compulsory: No Categories and Units details: Multiple choice: PVI, anterior wall, posterior wall, superior wall

      Variable: fluoro_time Display name: Time duration of fluoroscopy Type: Ablation Compulsory: No Categories and Units details: Minutes

      Variable: DLP Display name: Dose length product Type: Ablation Compulsory: No Categories and Units details: mGy*cm

      Variable: dwell_time Display name: Time in the left atrium (dwell time) Type: Ablation Compulsory: No Categories and Units details: Minutes; Defined as time since the catheters entered left atrium

      Variable: complications Display name: Complications during ablation Type: Ablation Compulsory: No Categories and Units details: if any, indicate what kind

ELIGIBILITY:
Inclusion Criteria:

- All patients with AF or AFl in whom TEE will be performed (to assess their eligibility for cardioversion or ablation), hospitalized in a participating center during study period (all consecutive patients).

Exclusion Criteria:

Age<18, lack of informed, written consent to the TEE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AF or AFl in whom TEE will be performed (to assess their eligibility for cardioversion or ablation), hospitalized in a participating center during study period.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of the presence of left atrial appendage thrombus in patients with atrial fibrillation or atrial flutter, in whom tranesophageal is performed before cardioversion or catheter ablation ablation. | One day
  We will asses the left atrial appendage in transesophageal echocardiography (TEEO for the presence of the left atrial appendage thrombus. During TEE we will record multiple projections of the left atrial appendage and we will measure laeft atrial appendage flows as listed below:
  1. Projection on LAA (Left Atrial Appendage): 0, 45, 90, 135 degrees, and other projections that are necessary to correctly image the entire LAA according to the investigator/ echocardiographer.
  2. 3D acquisition of the volume that contains LAA (multi-beat-optimized).
  3. Measurement of maximum emptying velocity of LAA 1cm from the LAA ostium - at least three measurements in two different scanning angles, averaged.
  4. Acquisition of spectral Doppler image of LAA emptying (three images from two or more scanning angles) (still images).

SECONDARY OUTCOMES:
Follow up for adverse outcomes | 1 year
  Follow-up for death, stroke, myocardial infarction, new onset or worsening of heart failure or acute limb ischemia. This will be obtained trough telephone interview.
Follow up for ablation recurrence | 1 year
  If possible, we will follow up the patients for AF recurrence.

OTHER OUTCOMES:
Electroanatomical data | One Day
  In patients who undergo catheter ablation with elepctroanatomical mapping we will collect and analyze data acquired during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Pieszko, MD, PhD, Principal Investigator — University of Zielona Gora
Locations (7):
- St. Anne Hospital, Brno, Czechia
- Poland (6):
  - Nowa Sol Multidyscyplinary Hospital, Nowa Sól, Lubusz Voivodeship
  - Medical University of Silesia, Katowice
  - John Paul II Hospital, Krakow
  - Military Institute of Medicine National Research Institute, Warsaw
  - National Institute of Cardiology, Warsaw
  - Collegium Medicum, University of Zielona Góra, Zielona Góra

IPD SHARING:
Plan to Share IPD: Yes
We plan to release an anonymized dataset in a public repository at the end of the study. This is depending on data sharing agreements with individual sites so the final dataset may not include all participating sites or all variables.
Supporting Information: Analytic Code
Time Frame: About 1 year after completion of the study.